CLINICAL TRIAL: NCT03094325
Title: On-pump Intraoperative Echocardiography (OPIE)
Brief Title: On-pump Intraoperative Echocardiography
Acronym: OPIE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 16-01729
Record Dates: First submitted 2017-03-23; First posted 2017-03-29 (Actual); Results first posted 2020-03-31 (Actual); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Septal Myectomy
Keywords: Septal Myectomy
MeSH Terms: interventions — Echocardiography, Transesophageal; Diagnostic Imaging

STUDY DESIGN:
Masking Description: Each of the 10 patients will have 4 measurements(OPIE & TEE before cardiopulmonary bypass and OPIE & TEE after cardiopulmonary bypass) in the septum using two techniques (TEE and OPIE Ultrasound Probe).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Septal myectomy (Experimental)
  Interventions: Device: Pre Operative On-pump intraoperative echocardiography; Device: Pre Operative Transesophageal echocardiography (TEE) imaging; Device: Post Operative On-pump intraoperative echocardiography; Device: Post Operative Transesophageal echocardiography (TEE) imaging

INTERVENTIONS:
Device: Pre Operative On-pump intraoperative echocardiography — Center tendency parameters(mean, standard deviation) will be reported for each outcome.
  Other Names: OPIE
Device: Pre Operative Transesophageal echocardiography (TEE) imaging — Center tendency parameters(mean, standard deviation) will be reported for each outcome.
  Other Names: TEE
Device: Post Operative On-pump intraoperative echocardiography — Center tendency parameters(mean, standard deviation) will be reported for each outcome.
Device: Post Operative Transesophageal echocardiography (TEE) imaging — Center tendency parameters(mean, standard deviation) will be reported for each outcome.

SUMMARY:
This pilot study uses an ultrasound probe that is currently clinically used to assess pituitary anatomy, the Hitachi-Aloka high resolution pituitary transducer to measure left ventricular (LV) septal thickness during cardiopulmonary bypass in the performance of surgical septal myectomy. Septal thickness will be assessed and can be visualized during the procedure and if it is likely to improve the efficacy and safety of the procedure. The probe has FDA clearance for a variety of intra-operative surgical procedures but will be off-label for this cardiac surgical protocol.

ELIGIBILITY:
Inclusion Criteria:

* scheduled to receive a septal myectomy.

Exclusion Criteria:

* Less than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-03-23 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-11-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Swistel, Principal Investigator — New York University Medical Center Institutional Review Boards
Locations (1):
- New York University School of Medicine, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All patients, inclusive of male and female and all racial/ethnic origins, age 18 or older who are scheduled to receive a septal myectomy
Groups:
- All Partcipants: Each of the 10 patients will have 4 measurements(OPIE & TEE before cardiopulmonary bypass and OPIE & TEE after cardiopulmonary bypass) in the septum using two techniques (TEE and OPIE Ultrasound Probe).
Period: Overall Study
Arm/Group | All Partcipants
Started | 10
TEE Before Cardiopulmonary Bypass | 10
OPIE Before Cardiopulmonary Bypass | 10
TEE After Cardiopulmonary Bypass | 10
OPIE After Cardiopulmonary Bypass | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Septal Myectomy
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Septal Thickness Measured Before Cardiopulmonary Bypass
Description: Center tendency parameters(mean, standard deviation)
Time Frame: 1 Day
Measure: Mean (Standard Deviation); unit: millimeters
Groups:
- TEE Measured Septal Thickness Before Cardiopulmonary Bypass: Post Operative Transesophageal echocardiography (TEE) imaging: Center tendency parameters(mean, standard deviation) will be reported for each outcome.
- OPIE Measured Thickness Before Cardiopulmonary Bypass: Post Operative On-pump intraoperative echocardiography: Center tendency parameters(mean, standard deviation) will be reported for each outcome
Arm/Group | TEE Measured Septal Thickness Before Cardiopulmonary Bypass | OPIE Measured Thickness Before Cardiopulmonary Bypass
Number analyzed (Participants) | 10 | 10
millimeters | 22.9 (4.6) | 22.5 (3.5)

ADVERSE EVENTS:
Time Frame: 1 year after cardiopulmonary bypass procedure
Arm/Group | TEE Measured Septal Thickness Before Cardiopulmonary Bypass | OPIE Measured Thickness Before Cardiopulmonary Bypass
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-06): https://cdn.clinicaltrials.gov/large-docs/25/NCT03094325/Prot_SAP_000.pdf